CLINICAL TRIAL: NCT05249335
Title: Comparison for Efficacy and Safety of Bowel Preparation Between Oral Sulfate Table and 2L-polyethylene Glycol/Ascorbate in Elderly: Multicenter, Prospective, Investigator Single-blinded, Randomized Study
Brief Title: Comparison for Efficacy and Safety of Bowel Preparation Between Oral Sulfate Table and 2L-polyethylene Glycol/Ascorbate in Elderly
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: unconfirmed yet
Record Dates: First submitted 2022-01-03; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-12

CONDITIONS: Colonic Disease; Intestinal Disease
Keywords: colonoscopy; orafang; bowel cleaning
MeSH Terms: conditions — Colonic Diseases; Intestinal Diseases

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, investigator single-blinded, randomized study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OST (Experimental): 2 days split dosing regimen
  Interventions: Drug: OST
- 2L-PEG/Asc (Active Comparator): 2 days split dosing regimen
  Interventions: Drug: 2L-PEG/Asc

INTERVENTIONS:
Drug: OST — The subject will receive Orafang for colonoscopy
  Arms: OST
Drug: 2L-PEG/Asc — The subject will receive 2L-PEG/Asc for colonoscopy
  Arms: 2L-PEG/Asc

SUMMARY:
This study compares the effectiveness and stability of intestinal tablet (OST), an oral sulfate table (OST), developed in the form of pills, with 2L-PEG/Asc for examinees aged 70 or older who are scheduled for colonoscopy.

DETAILED DESCRIPTION:
This study is comparison for efficacy and safety of bowel preparation between oral sulfate table and 2L-polyethylene glycol/ascorbate in elderly: multicenter, prospective, investigator single-blinded, randomized study. A total of 256 subjects will participate to this study and be assigned to the test group or the control group. The subject will administer the first dose of assigned investigational product in the evening prior to the scheduled colonoscopy. Subject will take the second dose early in the morning of the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age over 70
* Patients who is scheduled a colonoscopy
* Patients who is informed and give a consent in voluntary

Exclusion Criteria:

* History of colectomy
* Patients over American Society of Anesthesiology class III
* Patients who has difficulty swallowing
* In the case of abnormal findings requiring treatment in the basic blood test
* Patients with uncontrollable chronic diseases
* Patients suspected of having Paralytic ileus or intestinal obstruction.
* Patients who complains of alarm sign (severe abdominal pain, weight loss, anemia, gastrointestinal bleeding, etc.)
* Patients who has a history of drug abuse and addiction
* Patients who for any reason, are deemed by the Investigator to be inappropriate for this study

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Successful cleaning rate1 | Two days (from day of first dosing to day of colonoscopy)
  %Patient with Boston Bowel Preparation Scale (BBPS) scored over 2 in all segment
Successful cleaning rate2 | Two days (from day of first dosing to day of colonoscopy)
  %Patient with HCS-graded A or B

SECONDARY OUTCOMES:
Treatment compliance | Two days (from day of first dosing to day of colonoscopy)
  %Patient who have completed taking the investigational products

OTHER OUTCOMES:
Patient satisfaction assessed by questionnaire | Two days (from day of first dosing to day of colonoscopy)
  maximum score 10, minimum score0 , higher scores mean a better satisfaction
Adenoma/Polyp detection rate, ADR /PDR | Two days (from day of first dosing to day of colonoscopy)
  Adenoma/Polyp detection rate over 25%
clean cecal intubation time, colonoscopy time | Two days (from day of first dosing to day of colonoscopy)
  clean cecal intubation time, colonoscopy time

CONTACTS AND LOCATIONS:
Overall Officials: Cha Jaemyeong, M.D, Ph.D, Study Chair — Kyung Hee University Hospital at Gangdong; Gang Hoseok, M.D, Ph.D, Principal Investigator — HALLYM UNIV. MEDICAL CENTER; Seo Geomseok, M.D, Ph.D, Principal Investigator — Wonkwang University Hospital; Jeong Yunho, M.D, Ph.D, Principal Investigator — Soon Chun Hanyang University College of Medicine; Na Suyeong, M.D, Ph.D, Principal Investigator — Incheon St.Mary's Hospital

REFERENCES:
- [Derived] Kang HS, Na SY, Yoon JY, Jung Y, Seo GS, Cha JM. Efficacy, tolerability, and safety of oral sulfate tablet versus 2 L-polyethylene glycol/ascorbate for bowel preparation in older patients: prospective, multicenter, investigator single-blinded, randomized study. J Gastroenterol. 2024 May;59(5):402-410. doi: 10.1007/s00535-024-02089-9. Epub 2024 Mar 16. PMID 38492010